CLINICAL TRIAL: NCT02530216
Title: Automated Evaluation of Gastrointestinal Symptoms (AEGIS): A Pragmatic Clinical Trial Evaluating the Impact of AEGIS on Clinical Outcomes
Brief Title: Evaluating the Impact of Automated Evaluation of Gastrointestinal Symptoms (AEGIS) on Clinical Outcomes
Acronym: AEGIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Christopher Almario, Staff Physician and Health Services Research Scientist, Cedars-Sinai Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Pro00045243
Record Dates: First submitted 2015-08-19; First posted 2015-08-20 (Estimated); Last update posted 2018-05-01 (Actual); Status verified 2018-04

CONDITIONS: Abdominal Pain; Deglutition Disorders; Fecal Incontinence; Nausea; Diarrhea; Constipation; Gastroesophageal Reflux
MeSH Terms: conditions — Abdominal Pain; Deglutition Disorders; Fecal Incontinence; Nausea; Diarrhea; Constipation; Gastroesophageal Reflux

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual care (No Intervention): Individuals in this arm will undergo usual care with their physician.
- AEGIS (Automated Evaluation of Gastrointestinal Symptoms) (Experimental): Individuals in the AEGIS arm will be invited to use AEGIS/My GI Health prior to their clinic visit. For those who complete AEGIS/My GI Health, their physician will have access to their AEGIS symptom report (includes a GI symptom heat map and GI history) and tailored education prescription.
  Interventions: Other: AEGIS (Automated Evaluation of Gastrointestinal Symptoms)

INTERVENTIONS:
Other: AEGIS (Automated Evaluation of Gastrointestinal Symptoms) — AEGIS (Automated Evaluation of Gastrointestinal Symptoms) guides patients through questionnaires to measure symptom attributes including the timing, severity, frequency, location, quality, and character of their gastrointestinal (GI) symptoms, along with relevant comorbidities, family history, and alarm features. This information is transformed into a history of present illness (HPI) written in language familiar to clinicians. AEGIS also supports both the clinician and patient with an individualized "education prescription" which guides the patient through a library of multi-media educational materials on GI symptoms, conditions, and treatments. The prescription is created by the portal based on each patient's unique AEGIS "fingerprint."
  Arms: AEGIS (Automated Evaluation of Gastrointestinal Symptoms)

SUMMARY:
Healthcare delivery now mandates shorter visits with higher documentation requirements, undermining the patient-provider interaction. Electronic health records (EHRs) have the potential to improve outcomes and quality of care in this pressured environment, and are endorsed by the Patient Protection and Affordable Care Act (ACA) and Health Information Technology for Economic and Clinical Health (HITECH) Act as an important mechanism to support value-based healthcare. However, EHR systems were principally designed to support the transactional needs of administrators and billers, less so to nurture the relationship between patients and their providers. The purpose of this research is to identify ways to use EHRs to support clinical gastroenterologists and their patients while meeting the meaningful use requirements of the HITECH Act.

To improve clinic visit efficiency and meet criteria for meaningful use, investigators developed a patient-provider portal (P3) that systematically collects patient symptoms using a computer algorithm called Automated Evaluation of Gastrointestinal Symptoms (AEGIS). AEGIS utilizes computerized adaptive testing (CAT) to guide patients through questions drawn from a library of over 300 symptom attributes measuring the timing, severity, frequency, location, quality, and character of their GI symptoms, along with relevant comorbidities, family history, and alarm features. The system then automatically "translates" the patient report into a full narrative HPI available for use by GI providers in an EHR.

In a cross-sectional study in the American Journal of Gastroenterology comparing AEGIS versus physician-documented HPIs, investigators found that blinded physician reviewers perceived that AEGIS HPIs were of higher overall quality, better organized, and more succinct, comprehensible, complete and useful compared to HPIs written by physicians during usual care in academic GI clinics. In the current study, investigators aim to evaluate computer-generated HPIs prospectively on a wider scale in diverse academic and community-based settings. Moreover, investigators aim to test an enhanced AEGIS intervention that ties patient HPIs to an individualized "education prescription" which guides the patient through a library of multi-media educational materials on GI symptoms, conditions, and treatments.

ELIGIBILITY:
Inclusion Criteria:

* Presenting to the gastrointestinal clinic for evaluation.
* Able to read and write English.
* Has basic computing skills.

Exclusion Criteria:

* Having been seen and evaluated in the gastrointestinal clinic within the last 8 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 610 (Actual)
Dates: Start 2017-04-10 (Actual); Primary Completion 2018-02-07 (Actual); Study Completion 2018-02-07 (Actual)

PRIMARY OUTCOMES:
Prevalence of documented alarm symptoms | Completed and documented by the physician in the clinic note within 1 week of the initial clinic visit
  Prevalence of documented alarm symptoms (blood in the stool, unintentional weight loss, hematochezia, hematemesis) in the clinic note as documented by physicians.

SECONDARY OUTCOMES:
Prevalence of diagnosed organic disease | Organic disease (e.g., Celiac disease, inflammatory bowel disease, etc.) diagnosed within 6 months of the initial clinic visit
Time to diagnosis of organic disease | Time to diagnosis of organic disease (e.g., Celiac disease, inflammatory bowel disease, etc.) within 6 months of the initial clinic visit

CONTACTS AND LOCATIONS:
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States